CLINICAL TRIAL: NCT03223623
Title: Investigations of Pathophysiology of Focal Hand Dystonia
Brief Title: Pathophysiology of Focal Hand Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 170126; 17-N-0126
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-05-25

CONDITIONS: Dystonia
Keywords: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FHD (Active Comparator): adults with Focal Hand Dystonia
  Interventions: Device: TMS; Device: MRI; Device: VASO Imaging
- Healthy Volunteer (Placebo Comparator): adult healthy volunteers
  Interventions: Device: TMS; Device: MRI; Device: VASO Imaging

INTERVENTIONS:
Device: TMS — Single pulse TMS, IPL-M1 Interaction, IPL-M1 Interaction, Inhibitory Theta Burst Protocol (cTBS)
Device: MRI — High-resolution MRI for anatomical reference; fMRI scan as per research fMRI protocol will be conducted under 3 conditions. 1. Rest 2. Voluntary activity 3. Motor imagery task.
Device: VASO Imaging — The voluntary activity condition will involve 4 tasks: a. individual tapping of two fingers (index and little), b. individual tapping of four fingers (index, middle, ring, and little; no thumb) interspaced with rest periods, c. individual tapping of all five fingers (index, middle, ring, little, and thumb) interspaced with rest periods and d. Alternating grasping or retraction of a rubber ball interspaced with rest periods.

SUMMARY:
Background:

Little is known about the problems in brain function in focal hand dystonia (FHD) or complex regional pain syndrome (CRPS) dystonia. It is unclear why some CRPS patients develop dystonia but others do not. Researchers want to learn which area of the brain is involved in CRPS dystonia compared with FHD.

Objectives:

To understand why people with CRPS develop dystonia, and if these reasons are different in people with FHD.

Eligibility:

Adults ages 18 - 70 with CRPS dystonia OR with CRPS without dystonia OR with FHD and Healthy volunteers of similar age.

Design:

Participants will be screened with physical exam, neurological exam, and medical history. They may give a urine sample and will answer questions.

Participants can have 4 - 5 outpatient visits or stay at the clinical center for approximately 5-6 days.

Participants will have MRI scans. They will lie on a table that slides in and out of a scanner that takes pictures of their brain. They will do small tasks or be asked to imagine things during the scanning.

Participants will have transcranial magnetic stimulation (TMS) sessions for a few hours, with breaks. A brief electrical current passing through a well insulated wire coil on the scalp creates a magnetic pulse. This affects brain activity. Participants may do small tasks during TMS.

Participants will have the electrical activity of their muscles measured during TMS sessions. Small sticky pads will be attached to their hands and arms.

Participants ability to feel 2 separate stimuli as different will be tested by using a weak electrical shock to their fingers. They will also be asked to feel small plastic domes with ridges, that may cause discomfort.

DETAILED DESCRIPTION:
Objective: detailed evaluation of pathophysiology of Focal Hand Dystonia (FHD) with focus on the involvement of the parietal area, and to investigate differences in cortical mapping in the sensory and motor cortices between FHD and healthy volunteers.

Study population: The study will enroll patients with FHD and Healthy Volunteers (HVs).

Design: Prospective study using MRI and Physiology experiments using EMG and TMS based protocols to evaluate the differences between the groups.

Outcome measures: The evaluation using fMRI will be performed under 3 conditions; 1. Rest 2. Voluntary activity 3. Motor imagery task.

Outcome measures (fMRI based):

We will explore the differences in BOLD signal in the parietal lobe, in FHD compared to HVs, in the different conditions. We will look for changes in the BOLD signal in the parietal sensorimotor integration area.

We will use vascular occupancy imaging (VASO) to explore differences of detailed cortical mapping of neural structures between FHD and healthy volunteers.

The Physiology experiments aim to explore abnormalities and differences in the baseline motor cortical excitability between the groups and evaluate the influence of continuous Theta Burst Stimulation (cTBS) on these measures. We will study the influence of cTBS on the phenomenon Cortical Silent Period (cSP) in FHD.

We will also be studying the baseline Spatial and Temporal Discrimination (SDTs and TDTs), which are measures of sensory surround inhibition and have been noted to be endophenotypic of dystonia.

Physiology outcomes:

Baseline differential influences of PMv and IPL on motor cortical excitability and changes after cTBS of dIPL.

Baseline cortical Silent Period (cSP) in the involved and uninvolved limb in FHD and the influence of cTBS on cSP in the involved limb.

The TDTs/ SDTs in both the involved and uninvolved limbs in FHD compared to HVs.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy research volunteers and adult patients with FHD will be eligible for the study.

* Age between 18 - 70 years.
* Able to give informed consent.
* Able to comply with all study procedures.
* Subjects must be willing to abstain from alcohol for at least 48 hours prior to the study.
* Adult patients with an established diagnosis of FHD.
* Healthy volunteers will be healthy subjects without neurological or psychiatric disorders established by history and physical/neurological examination.
* Patients receiving botulinum toxin injections will be evaluated after 3 months since their last injection.
* All participants must be able to obtain an MRI (No contraindications per MRI safety checklist) which will be part of the initial evaluation.

EXCLUSION CRITERIA:

* Self-reported consumption of >14 alcoholic drinks/week for a man and >7 alcoholic drinks/week for a woman.
* Patients on daily chronic opioid or benzodiazepine use.
* Patients treated with anticholinergics, who are not willing and/or unable to withhold taking them for 1 week prior and for the duration of the study participation.
* Patients taking opioids and/or benzodiazepines on an as needed basis, who are not willing and/or unable to withhold taking them for 1 week or time interval equivalent to 5 half-lives (whichever is shorter) prior to study participation and for the days during study participation.
* Abnormal findings on neurological examination including cognitive impairment, except diagnosis of FHD in patients.
* History of or current brain tumor, stroke, head trauma with loss of consciousness, epilepsy or seizures.
* Past or present medical history of (a) neurological disorders, such as stroke, movement disorders (other than dystonia in the patient group), ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug dependence; (B) ventricular arrhythmias, renal and hepatic insufficiency, vascular headache, or carcinoid syndrome.
* Subjects with Baclofen pumps and/or neuro stimulators for pain.
* Current episode of major depression or any major psychiatric illness. Note: SSRI use is not exclusionary.
* Pregnant or breastfeeding women. Aside from history obtained at the screening, pregnancy status in women with childbearing potential is also established by urine pregnancy testing no more than 24 hours before each MRI and TMS sessions.
* Subjects who have contraindications to MRI:

  * You have metal in your body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if you were a welder or metal worker, since you may small metal fragments in the eye.
  * You are uncomfortable in small closed spaces (you have claustrophobia) so that you would feel uncomfortable in the MRI machine.
  * You are not able to lie comfortably on your back for approximately 2 hours.
* Subjects who have contra-indications for TMS

  * You have a pacemaker, implanted pump, stimulator, cochlear implant or metal objects inside the eye or skull.
  * You have hearing loss (assessed by participant self-report or history).
  * You are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
explore the differences in BOLD signal in the parietal lobe, in FHD compared to HVs, in the different conditions. | throughout
  We will look for changes in the BOLD signal in the parietal sensorimotor integration area.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.The anatomical MRI images obtained under this protocol will be made available to other NIH investigators on PACS (radlite.cc.nih.gov) or the NMR (oxygen.nimh.nih.gov) data server for sharing with other NIH protocols immediately after acquisition. @@@@@@All de-identified data will be shared at the time of publication or later using the NINDS data repository (data.ninds.nih.gov). Data that may be shared with investigators outside NIH will be reported at the time of Continuing Review. Submissions to NIH-sponsored or supported databases and repositories will be reported at the time of Continuing Review. Submission to non-NIH sponsored or supported databases and repositories will be submitted for prospective IRB approval.
Supporting Information: Study Protocol
Time Frame: anatomical MRI images to other NIH investigators: upon acquisition.@@@@@@All de-identified data: 6 months after publication.
Access Criteria: The anatomical MRI images obtained under this protocol will be made available to other NIH investigators on PACS (radlite.cc.nih.gov) or the NMR (oxygen.nimh.nih.gov) data server for sharing with other NIH protocols immediately after acquisition. @@@@@@All de-identified data will be shared at the time of publication or later using the NINDS data repository (data.ninds.nih.gov). Data that may be shared with investigators outside NIH will be reported at the time of Continuing Review. Submissions to NIH-sponsored or supported databases and repositories will be reported at the time of Continuing Review. Submission to non-NIH sponsored or supported databases and repositories will be submitted for prospective IRB approval.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-N-0126.html